CLINICAL TRIAL: NCT01417078
Title: An Open-Label Study to Determine the Pharmacokinetics of a Single Dose of Diazepam Nasal Spray in Adult Epileptic Patients Experiencing a Seizure Episode for Which Acute Treatment With a Benzodiazepine is Clinically Indicated
Brief Title: A Pharmacokinetic Study of a Single-Dose of Diazepam Nasal Spray in Adult Epileptic Patients Experiencing a Seizure Episode
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZNS-ARS-103
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diazepam Nasal Spray (Experimental)
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — single-dose; dosage in mg, based on patient body weight

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of Diazepam Nasal Spray following a single dose in epileptic patients experiencing a seizure episode.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent for study participation.
* General good health with no clinically significant unstable abnormalities.
* Diagnosis of epilepsy.

Exclusion Criteria:

* Individuals receiving warfarin (Coumadin®) or dabigatran (Pradaxa®).
* Use of any investigational drug within 30 days.
* Blood or plasma donation within 30 days.
* Not willing or unable to tolerate blood draws.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Ward, MD, Study Director — Neuronex, Inc.
Locations (4):
- United States (4):
  - Barrow Neurology Clinics at St Joseph's Hospital, Phoenix, Arizona
  - Johns Hopkins University, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diazepam Nasal Spray
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Population Number (N)=31 Pharmacokinetic Population N=30
Arm/Group | Diazepam Nasal Spray
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2)] | 26.3 (4.08)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Measure Plasma Concentration (Cmax),
Description: Summary of Dose-Adjusted Diazepam and Nordiazepam PK parameter Cmax. The mean Cmax value was adjusted to a 20 mg dose.
Time Frame: Pre-dose, 10, 15, 30, and 45 mins, and 1, 1.5, 2, 4, 6, 9,and 12 hours
Population: PK Population: patients who had adequate concentration-time data to permit estimation of noncompartmental PK parameters.
  One patient was not included in the analysis of nordiazepam due to receiving clorazepate, which interfered with the analysis of nordiazepam from diazepam administration.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Groups:
- Nordiazepam: Diazepam was slowly converted to nordiazepam following intranasal administration
Arm/Group | Diazepam Nasal Spray | Nordiazepam
Number analyzed (Participants) | 30 | 29
nanogram/milliliter (ng/mL) | 208 (90.3) | 23.9 (16.5)

2. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs refer to adverse events with start dates occurring after dosing. Treatment-Related TEAEs refer to those 'possibly' or 'probably' related to study drug.
  Intensity definitions:
  * Mild: Usually transient, required no special treatment, and did not interfere with the patient's daily activities.
  * Moderate: Usually caused a low degree of inconvenience or concern to the patient, and may have interfered with daily activities, but was usually ameliorated by simple therapeutic measures.
  * Severe: Interrupted a patient's usual daily activities, and generally required systemic drug therapy or other treatment.
Time Frame: Pre-dose to 48 hours post-dose
Population: Safety Population (dosed with study drug)
Measure: Number; unit: participants
Arm/Group | Diazepam Nasal Spray
Number analyzed (Participants) | 31
participants
  Subjects with one or more TEAEs | 28
  Total number of TEAEs | 96
  Subjects with one or more Treatment-Related TEAEs | 21
  Total number of Treatment-Related TEAEs | 56
  Subjects with one or more Severe TEAEs | 1
  Total number of Severe TEAEs | 1
  Total number of Moderate TEAEs | 24
  Total number of Mild TEAEs | 71

3. Primary Outcome: Pharmacokinetic (PK) Parameter: Time to Maximum Plasma Concentration (Tmax)
Description: Summary of Dose-Adjusted Diazepam and Nordiazepam PK parameter Tmax.
  The mean Tmax value was adjusted to a 20 mg dose.
Time Frame: Pre-dose, 10, 15, 30, and 45 mins, and 1, 1.5, 2, 4, 6, 9,and 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Diazepam Nasal Spray | Nordiazepam
Number analyzed (Participants) | 30 | 29
hour (h) | 0.98 (0.86) | 11.10 (2.14)

4. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under The Concentration Curve From Time 0 to 12 Hours (AUC(0-12)) and AUC Time to Last Measurable Plasma Concentration
Description: Summary of Dose-Adjusted Diazepam and Nordiazepam PK parameter AUC(0-12) and AUC(last).
  The mean estimate of AUC(0-12) was adjusted to a 20 mg dose. AUC(last) was used for the calculation of AUC for nordiazepam. AUC(0-12) values could not be estimated for nordiazepam given that nordiazepam concentrations were rising between 6 and 12 hours.
Time Frame: Pre-dose, 10, 15, 30, and 45 mins, and 1, 1.5, 2, 4, 6, 9,and 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Diazepam Nasal Spray | Nordiazepam
Number analyzed (Participants) | 30 | 29
hour*nanogram/milliliter (h*ng/mL)
  AUC(0-12) | 1227 (488) | NA (NA) — AUC(0-12) values could not be estimated for nordiazepam given that nordiazepam concentrations were rising between 6 and 12 hours
  AUC(last) | NA (NA) — AUC(last) was used for the calculation of AUC for nordiazepam. | 192 (148)

ADVERSE EVENTS:
Time Frame: Pre-dose to 48 hours post-dose
Description: TEAEs refer to AEs with start date and times occuring after dosing.
Arm/Group | Diazepam Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 28/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diazepam Nasal Spray (N=31)
Headache (Nervous system disorders) | 16
Dysgeusia (Nervous system disorders) | 8
Somnolence (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Parosmia (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 1
Lacrimation increased (Eye disorders) | 5
Fatigue (General disorders) | 2
Catheter site pain (General disorders) | 1
Feeling hot (General disorders) | 1
Peripheral coldness (General disorders) | 1
Tongue injury (Injury, poisoning and procedural complications) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Blood pressure increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Urinary retention (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has right to review at least forty-five (45) days prior to the date of submission for publication or of public disclosure. Multi-center trials; publication shall be delayed until a publication of the multi-center results or until twelve (12) months have elapsed since the completion of the study, whichever occurs first.